CLINICAL TRIAL: NCT04919252
Title: Efficacy and Safety of Vedolizumab in Biologic-naïve Korean Patients With Moderate to Severe Inflammatory Bowel Disease
Acronym: VEDOKO-IIT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2020-1365
Record Dates: First submitted 2021-04-06; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Crohn's Disease and Ulcerative Colitis
Keywords: inflammatory bowel disease
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vedolizumab (Experimental): * Crohn's disease (CD): If a subject does not respond to vedolizumab 300mg iv 0, 2, and 6 weeks for induction, an additional dose of vedolizumab 300 mg will be given at week 10. On the other hand, Maintenance therapy should be continued every 8 weeks from week 14 in responding patients, and for some patients who have experienced a decrease in their response, it can be given every 4 weeks. The maximum dosing period is 54 weeks.
  * Ulcerative colitis (UC): If a subject responds to vedolizumab 300mg iv 0, 2, and 6 weeks for induction, maintenance therapy should be continued every 8 weeks from week 14, and for some patients who have experienced a decrease in their response, it can be given every 4 weeks. The maximum dosing period is 54 weeks.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — * Crohn's disease (CD): If a subject does not respond to vedolizumab 300mg iv 0, 2, and 6 weeks for induction, an additional dose of vedolizumab 300 mg will be given at week 10. On the other hand, Maintenance therapy should be continued every 8 weeks from week 14 in responding patients, and for some patients who have experienced a decrease in their response, it can be given every 4 weeks. The maximum dosing period is 54 weeks.
  * Ulcerative colitis (UC): If a subject responds to vedolizumab 300mg iv 0, 2, and 6 weeks for induction, maintenance therapy should be continued every 8 weeks from week 14, and for some patients who have experienced a decrease in their response, it can be given every 4 weeks. The maximum dosing period is 54 weeks.

SUMMARY:
If subjects voluntarily consent to participation in the study, those who are finally determined to be eligible for the study after whether all of the inclusion criteria and none of the exclusion criteria are met is checked will receive the study drug. Efficacy and safety will be evaluated at baseline, baseline, 2 weeks, 6 weeks, 14 weeks, 22 weeks, 30 weeks, 38 weeks, 46 weeks, and 54 weeks.

DETAILED DESCRIPTION:
This study, which is designed as a multicenter, open-label, single-arm, phase 3b clinical trial, is intended to evaluate the efficacy and safety of vedolizumab in biologic-naïve Korean patients with moderate-to-severe bowel disease.

The study is conducted with a single arm, and the subjects to be recruited consist of 30 patients with Crohn's disease and 30 patients with ulcerative colitis (considering dropout rate of 20%).

The total period after the subject enrollment is 54 weeks, and a total of 10 visits are made with screening, baseline, 2 weeks, 6 weeks, 14 weeks, 22 weeks, 30 weeks, 38 weeks, 46 weeks, and 54 weeks.

* Crohn's disease (CD): If a subject does not respond to vedolizumab 300mg iv 0, 2, and 6 weeks for induction, an additional dose of vedolizumab 300 mg will be given at week 10. On the other hand, Maintenance therapy should be continued every 8 weeks from week 14 in responding patients, and for some patients who have experienced a decrease in their response, it can be given every 4 weeks.The maximum dosing period is 54 weeks.
* Ulcerative colitis (UC): If a subject responds to vedolizumab 300mg iv 0, 2, and 6 weeks for induction, maintenance therapy should be continued every 8 weeks from week 14, and for some patients who have experienced a decrease in their response, it can be given every 4 weeks.The maximum dosing period is 54 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥ 19 years to ≤ 70 years
2. Patients with moderate-to-severe active Crohn's disease or ulcerative colitis who are unresponsive to, become unresponsive to, or have no tolerability to universal treatment (with corticosteroids, immunomodulators, etc.)

   * CDAI (Crohn's Disease Activity Index) ≥ 220 for Crohn's disease
   * Complete Mayo score ≥ 6 for ulcerative colitis

Exclusion Criteria:

1. A history of total colectomy
2. Acute severe UC(Ulcerative Colitis)
3. A potential for a bowel resection surgery within 3 months
4. Pregnancy and breastfeeding
5. Prior use of any biologics including anti-TNFs, ustekinumab, and tofacitinib
6. A history of solid cancer and blood cancer within 5 years
7. Positive for active or latent tuberculosis (However, screening is possible if active tuberculosis is excluded and after at least 4 weeks of latent tuberculosis treatment.)
8. Active severe infections such as sepsis, cytomegalovirus, listeriosis, and opportunistic infections such as progressive multifocal leukoencephalopathy (PML).
9. Hypersensitivity to vedolizumab or its substances (e.g., dyspnoea, bronchospasm, redness, and increased heart rate)
10. Experience of treatment with a drug or a medical device due to participation in another clinical trial within 3 months from the date of consent
11. A woman of childbearing potential who has a positive pregnancy test (Urine-hCG or Serum hCG) at a screening visit or does not agree to use at least one of medically acceptable, effective contraceptive methods*. However, females who reached menopause at least one year ago or turned out infertile due to an operation should be excluded.

    *Effective contraceptive methods: intrauterine devices (e.g., IUD, mirena), dual barrier methods (diaphragm or condom/femidom + spermicide), and parenteral contraceptives. Continuing only sexual abstinence is not viewed as an acceptable method.
12. A woman of childbearing potential who neither practices adequate contraception nor agrees to continue its use for at least 18 weeks after the last dose of the study drug.
13. Those decided by the investigator to be not eligible for this study

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Clinical remission rate (%) at 14 weeks after commencement of vedolizumab treatment in induction phase | 14 weeks
  Clinical remission is defined as Mayo score ≤ 2 points and individual score ≤ 1 point for Ulcerative colitis and CDAI(Crohn's Disease Activity Index) < 150 for Crohn's Disease.
Clinical remission rate (%) at 54 weeks in maintenance phase | 54 weeks
  Clinical remission is defined as Mayo score ≤ 2 points and individual score ≤ 1 point for Ulcerative colitis and CDAI(Crohn's Disease Activity Index) < 150 for Crohn's Disease.

SECONDARY OUTCOMES:
Response rate of dose intensification at 54 weeks in inadequate responders at 6 weeks | 6 weeks, 54 weeks
  Response rate of dose intensification at 54 weeks in inadequate responders at 6 weeks
Mucosal healing rate at 14 weeks and 54 weeks | 14 weeks, 54 weeks
  Mucosal healing is defined as Mayo endoscopic subscore ≤ 1 for UC and as no visible ulcer for Crohn's Disease.
Steroid free remission rate at 54 weeks | 54 weeks
  Steroid free remission rate at 54 weeks
Transmural healing rate at 14 weeks and 54 weeks for Crohn's Disease | 14 weeks, 54 weeks
  Transmural healing is defined as normal cross-sectional imaging and mucosal healing.
Correlation of CRP(C-reactive protein) level with clinical remission at 54 weeks. | 54 weeks
  The logistic regression will analyze CRP level to see the correlation with clinical remission.
Correlation of fecal calprotectin level with clinical remission at 54 weeks | 54 weeks
  The logistic regression will analyze fecal calprotectin level to see the correlation with clinical remission.
Correlation of endoscopic severity with clinical remission at 54 weeks | 54 weeks
  The logistic regression will analyze endoscopic severity to see the correlation with clinical remission.
Correlation of radiologic severity with clinical remission at 54 weeks | 54 weeks
  The quality of life(QoL) will be assessed by IBDQ(Inflammatory Bowel The logistic regression will analyze radiologic severity to see the correlation with clinical remission.
Correlation of CDAI(Crohn's Disease Activity Index) score with clinical remission at 54 weeks | 54 weeks
  The logistic regression will analyze CDAI score to see the correlation with clinical remission.
Correlation of Mayo score with clinical remission at 54 weeks | 54 weeks
  The logistic regression will analyze Mayo score to see the correlation with clinical remission.
Changes in fecal microbiota after vedolizumab treatment: Microbiota change will be compared with baseline status using α diversity and β diversity. | Baseline, 14 weeks, 54 weeks
  Changes in fecal microbiota at 14 weeks and 54 weeks after treatment versus baseline are evaluated by α-diversity and β-diversity.
QoL(Quality of Life): IBDQ(Inflammatory Bowel Disease Questionnaire) | Baseline, 14 weeks, 54 weeks
  The quality of life(QoL) will be assessed by IBDQ(Inflammatory Bowel Disease Questionnaire) survey at week 0, week 14 and week 54. A paired data analysis will be conducted at week 14 and week 54 compared to week 0 (before treatment). It will be evaluated in Crohn's Disease and Ulcerative colitis, separately.

CONTACTS AND LOCATIONS:
Overall Officials: Jae hee Cheon, MD, PhD, Principal Investigator — Severance Hospital of Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No